CLINICAL TRIAL: NCT03399110
Title: XELOX for 4 Months Versus 6 Months as Adjuvant Chemotherapy in Gastric Cancer After D2 Resection (LOMAC)
Brief Title: XELOX for 4 Months Versus 6 Months in Gastric Cancer (LOMAC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCGC005
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer,Adjuvant chemtherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XELOX for 4 months (Experimental): Adjuvant chemotherapy with capecitabine and oxaliplatin after surgery consists of 5 to 6 cycles, each lasting 3 weeks: oral capecitabine at 1000 mg/m² twice daily on days 1-14, combined with intravenous oxaliplatin at 130 mg/m² on day 1, administered for 5 to 6 months or until disease progression.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- XELOX for 6 months (Active Comparator): Adjuvant chemotherapy with capecitabine and oxaliplatin after surgery consists of eight 3-week cycles: oral capecitabine at 1000 mg/m² twice daily on days 1-14, combined with intravenous oxaliplatin at 130 mg/m² on day 1, administered for 6 months or until disease progression.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2
  Other Names: Eloxatin
Drug: Capecitabine — Capecitabine 1000mg/m2
  Other Names: Xeloda

SUMMARY:
Our study aims to compare the efficacy and safety of 4-month versus 6-month adjuvant chemotherapy with capecitabine and oxaliplatin following D2 gastrectomy in patients with gastric cancer.

Hypothesis: In patients with gastric cancer who have undergone D2 gastrectomy, a 4-month regimen of capecitabine and oxaliplatin demonstrates noninferiority to a 6-month regimen in terms of disease-free survival (DFS) and safety.

DETAILED DESCRIPTION:
Surgical resection is the cornerstone of treatment for patients with localized gastric cancer. In the CLASSIC trial, capecitabine plus oxaliplatin for 6 months following D2 gastrectomy has been established as an effective postoperative adjuvant treatment for patients with operable stage II or III gastric cancer. However, due to adverse events, chemotherapy discontinuations occurred in 50 (10%) patients, primarily due to nausea, neutropenia, decreased appetite, peripheral neuropathy, diarrhea, and vomiting. At the 2017 ASCO Annual Meeting, Grothey et al. reported the results of the IDEA trial. For patients with lymph node-positive colon cancer (stage III), some may benefit from a shorter duration of chemotherapy post-surgery. An analysis of six clinical trials involving over 12,800 patients showed that 3 months of chemotherapy was nearly as effective as 6 months for patients with a lower recurrence risk, while also causing fewer side effects, particularly nerve damage. Based on the findings from the IDEA trial, we hypothesize that a 4-month regimen of capecitabine plus oxaliplatin may also benefit patients following D2 gastrectomy while reducing adverse events compared with the standard 6-month regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Histologically confirmed primary adenocarcinoma of the stomach, staged as II, IIIA, or IIIB according to pathological findings.
3. R0 resection and D2 gastrectomy performed.
4. No other concurrent malignancies.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. No contraindications to chemotherapy.

Exclusion Criteria:

1. Receipt of preoperative treatment, including radiation therapy, chemotherapy, or immunotherapy.
2. Patients with stage I, IIIC, or IV gastric cancer.
3. Presence of severe organ diseases, including heart, lung, brain, liver, or other vital organ dysfunction.
4. Known or suspected drug allergies.
5. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
DFS | 3-year
  Disease-free survival

SECONDARY OUTCOMES:
Adverse Events | 6-month
  Adverse Events of Chemotherapy
OS | 3-year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD, MD, Principal Investigator — Fudan University
Locations (9):
- China (9):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei
  - Jiangsu Cancer Hospital, Nanjing
  - Changhai Hospital, Shanghai
  - Second Affiliated Hospital (Changzheng Hospital) of Naval Medical University, Shanghai
  - Shanghai East Hospital, Shanghai
  - 13940152108@163.Com, Shenyang
  - The First Affiliated Hospital of Wannan Medical College, Wuhu

IPD SHARING:
Plan to Share IPD: Undecided